Official Title: Infracalcaneal Peppering Injection Technique for Chronic Plantar Fasciitis: Protocol for a Parallel Randomized Clinical Trial

NCT05868577

IRB Approval Date: 04/05/2024

Study Title: Infracalcaneal Peppering Injection Technique for Chronic Plantar Fasciitis: Protocol for a Parallel Randomized Clinical Trial

Principal Investigator: Michael A. Jones, DPM, FACFAS
Atrium Health Wake Forest Baptist
Podiatry-Westchester
1814 Westchester Drive, Suite 300
High Point, NC 27262
michione@wakehealth.edu

Sub-Investigators: David W. Robinson, MD; David R. Sinacore, PT, PhD, FAPTA; Dekarlos M. Dial, DPM, FACFAS; Kerry A. Danelson, PhD; Garrett S. Bullock, PT, DPT, DPhil

**Sponsor or funding source: CTSI** 

### **Background, Rationale and Context**

Plantar fasciitis is one of the most common causes of foot pain in adults. Plantar fasciitis demonstrates a lifetime prevalence rate of 10% and accounts for 1 million provider visits in the United States annually (1). In 2007, an estimated \$284 million was spent on medical treatments for this condition (2).

Briefly, from an anatomical perspective, the plantar fascia is *not* inert. This thick band of tissue (*aponeurosis*) on the underside of the foot comprises three bands (i.e., medial, central, and lateral) that connect the calcaneus to the toes, has intimate involvement with the Achilles tendon, and acts as both a dynamic shock absorber as well a secondary support structure of the arch (3). As the toes extend during the stance phase of gait, the plantar fascia tightens, creating a *windlass mechanism* (4) that results in elevation of the foot arch, inversion of the hindfoot, and, consequently, external rotation of the leg. The plantar fascia is actually well innervated and together with the intrinsic foot musculature plays a *critical role* in both proprioception and stability, serves to stabilize the arch, and provides dynamic sensory and motor control to the foot (3). Thus, when the plantar fascia becomes irritated or *unhealthy*, this can have detrimental effects on an individual's ability for both standing and walking, which for most is *essential* for living. Unfortunately, the etiology of plantar fasciitis is still poorly understood despite numerous studies on this condition (5).

Thought to have primarily a *mechanical* origin, plantar fasciitis and its development is multifactorial, but *strongly associated* in individuals with an increased BMI (7) and/or decreased ankle joint dorsiflexion (i.e. calf muscle tightness) (8). The diagnosis of plantar fasciitis is usually based on *clinical criteria alone*, with pain localized to the medial tubercle of the calcaneus (i.e. its origin or *enthesis*) considered pathognomonic and is the most widely reported clinical sign. Most patients with plantar fasciitis report *plantar heel pain* after standing up from bed in the morning and/or after they have been seated for a prolonged time. Typically, the heel pain improves somewhat with ambulation but could intensify by day's end with prolonged walking or standing. Patients will oftentimes compensate with their gait to avoid placing direct pressure on the heel. Imaging plays a limited role in routine clinical practice, though may be useful to rule out other causes of heel pain when in doubt (6). As in other musculoskeletal disorders, plantar fasciitis has shown associations with increased levels of depression, stress, and anxiety and may have a significant negative impact on foot-specific and general health-related quality of life (9-10).

In terms of management, conservative therapy (e.g. stretching and/or strengthening exercises, self-myofascial release, NSAIDs, taping, arch supports, supportive shoes, rest, immobilization, etc. to name a few) is still viewed as the mainstay of treatment (11).

Protocol version: 7 Template updated 9.24.14 Interestingly, evidence on long-term prognosis of plantar fasciitis appears equivocal and no one treatment is superior to the others. Though most experts tout plantar fasciitis as a self-limiting condition (12), some *chronic* sufferers report continued issues with this disorder *5-15 years* from initial onset of symptoms (13), contributing to further ambivalence associated with this disorder. Surgery, typically performed by partially cutting the plantar fascia at the heel, can be offered in recalcitrant cases as a last resort. This *invasive* intervention is of course not without risks, including possible incomplete relief of symptoms (or, worse yet, *more pain* than before surgery), nerve damage, and permanent changes in foot shape (i.e. flat foot). Moreover, plantar fasciitis surgery in the US can cost \$10,000 or more (which varies by geography, surgeon's fees, facility costs, and other services such as anesthesia and follow up care) (14).

Lying within the conservative-surgical treatment spectrum for plantar fasciitis is local corticosteroid injection (CSI) therapy (15), a minimally invasive intervention that is relatively quick and easy for the clinician to perform in the outpatient clinical setting. A targeted plantar fascia injection typically combines both corticosteroid (CSI) and a local anesthetic (LA) as the substance infused (i.e. iniectate). Administration of a CSI near the irritated plantar fascia has documented evidence of providing pain relief for up to 1 month only (16). A randomized trial performed as far back as 1956 showed no statistical difference between CSI and placebo (i.e., saline) with 6-18 months of follow-up recorded (17). Yet, to this day, a CSI is essentially the only immediate intervention that can be proffered in the outpatient clinic by providers that thirdparty payers (at least in the United States) will compensate for. In point of fact, 73% of surveyed orthopaedic surgeons preferred CSI to treat heel pain (18), yet its own preeminent foot association, the American Orthopaedic Foot and Ankle Society (14), advocates for its judicious use for fear of deleterious side effects, including fat pad atrophy (20) and possible rupture (21). The ambiguity surrounding corticosteroid *injection* as therapy is further substantiated from histopathologic studies involving plantar fasciitis (22-24), which failed to demonstrate any inflammatory process, calling into question the rationale on the use of corticosteroids altogether, which are used primarily for their potent anti-inflammatory effects (18). Reasonably, the terminology plantar fasciitis is perhaps a misnomer given the degenerative (rather than inflammatory) findings uncovered (24), which some investigators refer to as plantar fasciosis or plantar fasciopathy, given the similar tissue pathology seen in other musculoskeletal tendon disorders, or tendinopathies (25-28, 31).

While there have been several prospective investigative studies on CSI for plantar fasciitis, there is vagueness on injection method. There are essentially two described techniques (29): single injection (how CSI is traditionally administered) or peppering injection, the latter initially described in 1964 (30) as a technique for lateral epicondylitis, a form of chronic tendinopathy involving the arm. Injection peppering is thought to disrupt the chronic degenerative process by provoking bleeding and inflammation to promote healing (31). Several study trials involving the injection method for lateral epicondylitis highlights that it is the physical needling of the pathologic site (i.e. peppering) as opposed to the injectate that incites healing (30-34). Thus, a peppering injection performed for plantar fasciitis, though just hypothetical, would act similarly via repeatedly fenestrating the pathologic site and opening holes on several spots rather than a single spot (33) to stimulate hematoma formation and subsequent healing. To our knowledge, only two previous investigative studies have disclosed its use for plantar fasciitis (35, 36). Likewise, the medical evidence on injection therapy for plantar fasciitis also shows imprecision on both the approach (i.e. medial or plantar heel) and target (i.e. superficial to, deep to, or into the plantar fascia) to inject, just as long as it is deposited close to the plantar fascia origin (enthesis) (19, 25, 37-39). Though ultrasound guidance can provide more realtime accuracy of where the injectate infiltrates, it shows no superiority to traditional palpation guided injection therapy (36).

Our research team considers corticosteroid injection a nebulous and insufficient treatment option for plantar fasciitis sufferers. If *first do no harm* is the physician's axiom, then

CSI's continued utilization altogether for this tricky pathology should be questioned. Our investigative team has exposed a knowledge gap and posits a challenge to the existing CSI treatment paradigm for plantar fasciitis via an alternative minimally invasive infracalcaneal peppering injection technique being non-inferior to traditional CSI, with the premise that it is the needle rather than the steroid administered that is beneficial for the patient.

Successful completion of our proposed pilot study addresses a critical knowledge gap in the treatment of chronic plantar fasciitis and breaches the translational roadblock of clinical implementation. The results from this rigorous pilot study will provide the framework for our anticipated full-scale efficacy trial with the potential of affording the clinician an upgraded evidenced-based treatment option that has been demonstrated to be safe, effective, and reproducible.

# **Objectives**

- 1. Assess feasibility of infracalcaneal peppering injection technique with and without CSI in the management of patients with chronic plantar fasciitis.
  - a. Feasibility of recruitment, randomization, retention, patient and physician time constraints, and tolerability of treatment will be assessed. Clear quantitative benchmarks and a number needed to treat will be achieved for planned utilization in a subsequent full-scale efficacy trial.
- 2. Assess the efficacy of infracalcaneal peppering injection with and without CSI for reduction in pain utilizing two validated patient reported outcomes measures (PROMs): the Visual Analog Scale (VAS) and Foot Function Index (FFI), administered at baseline, then at 2, 4, 8, and 12 weeks. Minimal Important Difference (MID) calculations for both VAS and FFI PROMs, specifically for plantar fasciitis, have already been investigated/established and will be used as a reference.
  - a. Greater than 75% of these PROMs from ALL cumulative target dates will be captured, providing a target number needed to treat (NNT) to conduct a full-scale efficacy trial investigation.

#### **Methods and Measures**

**Design:** A randomized, double-blind placebo-controlled pilot study at one single institution

**Setting:** Atrium Health Wake Forest Baptist Department of Orthopaedic Surgery-Podiatry Services practice located in High Point, North Carolina

### **Subject Selection Criteria**

#### **Inclusion Criteria**

- Men and women 18 years of age and older
- Patient reported history of plantar heel pain and confirmed clinical tenderness of pain with direct palpation of the medial calcaneal tubercle on baseline exam
- Diagnosis of chronic plantar fasciitis, defined for study purposes as symptoms greater than or equal to 6 weeks in duration

#### **Exclusion Criteria**

- Individuals less than 18 years of age
- Pregnancy

Protocol version: 7

- History of receiving a local heel injection (i.e. CSI or other injectate) within the last 3 months
- Prior heel trauma or surgery
- Allergy to local corticosteroid or local anesthesia

## **Sample Size**

We estimate the sample size required to answer the research question to be 50 participants.

#### **Interventions and Interactions**

Once both informed consent and enrollment have been verified, initial evaluation by the PI will be conducted on participants, and baseline assessments will be performed. The assessments include:

- Documentation of participant age at enrollment along with information on sex/gender, race, and ethnicity to ensure the study involves Inclusion of Individuals across the Lifespan
- History and physical exam
- Calculated BMI
- Documentation of referral patterns (PCP, self, or other referral)
  - If from PCP or other, documentation of what information/work-up was provided (e.g. told they have "heel spur", given NSAIDs, exercises, etc.)
- Clinical confirmation/diagnosis of plantar fasciitis (pain at medial calcaneal tubercle)
- Dolorimeter readings of PPT # (pressure algometer)
- Documentation of subjective reporting of first-step pain (yes/no)
- Foot posture score
- Heel tenderness score
- Initial X-ray (notation and measurement of heel spur) of the symptomatic foot/heel will be performed, if not already completed
- Initial diagnostic musculoskeletal US (PF thickness and echogenicity; fat pad thickness)
- Patient completed baseline self-assessment of both "general heel pain" and "first step pain" (VAS PROM)
- Patient completed baseline self-assessment of foot function (FFI PROM)

At this point, the patient will be block allocated to their study arm, having been randomized in a double-blind fashion by the clinical coordinator. This individual will facilitate safe record-keeping and the processes required to maintain the double-blind design of this study. We will specifically conduct the study in a permuted block design to ensure a 1:1 ratio for the two treatment intervention groups. The study arms are as follows:

- Group 1 CSI/LA injection
- Group 2 LA/Saline injection

A nurse or staff member will open a previously prepared and sealed opaque envelope (prepared beforehand by the clinical coordinator) labeled with the participant ID of the patient, which will be unique to the individual and different from their MRN. In this envelope, they will discover the patient's assigned treatment arm. The nurse or staff member will then prepare the syringe with the assigned treatment arm. Once the syringe is filled with the designated substance, the syringe will be wrapped with opaque tape or dark Coban wrap to conceal the contents in the

syringe for both the PI and study participant. The participant's skin will be sterilely prepped with alcohol.

The PI will then administer the injection using an infracalcaneal needle peppering technique as follows:

- 1. The hypodermic needle is inserted using infracalcaneal injection approach.
- 2. The hypodermic needle is withdrawn while at the same depositing injectate.
- 3. The hypodermic needle is redirected without emerging from the skin.

The PI will perform steps 1-3 standardly 20-25 times. Following the completion of the injection and clinical observation, the patient will receive home care and follow-up instructions which will include the standardized teaching of 3 exercises (calf stretching, plantar fascia specific stretching, and plantar fascia loading exercise). Patients will be sent home with an exercise diary to record when and if they complete the instructed exercises with directions to bring the diary to the next visit. Patients will receive 1 phone call between this visit and the next to check in on their exercise progress and remind them to complete the exercise diary.

The patient will be seen at follow-up visit #1 for evaluation and management 2 weeks post-treatment intervention. At this visit, the following assessments will be completed:

- History and physical exam
- Patient self-assessment of both "general heel pain" and "first step pain" (VAS PROM)
- Patient self-assessment of foot function (FFI PROM)
- Dolorimeter readings of PPT # (pressure algometer)
- Heel tenderness score
- Review of the exercise diary

A new exercise diary will be given to the patient. The recommended exercises will be instructed again. Patients will be encouraged to bring the diary to their next visit. To increase compliance, patients will receive 1 phone call to check in on their exercise progress and remind them to complete the exercise diary.

The patient will return for follow-up visit #2 for evaluation and management 4 weeks post-treatment intervention. At this visit, the following assessments will be completed:

- History and physical exam
- Patient self-assessment of both "general heel pain" and "first step pain" (VAS PROM)
- Patient self-assessment of foot function (FFI PROM)
- Dolorimeter readings of PPT # (pressure algometer)
- Heel tenderness score
- Review of the exercise diary

A new exercise diary will be given to the patient. The recommended exercises will be instructed again. Patients will be encouraged to bring the diary to their next visit. The patient will be called 1 time to remind them to complete their exercise diary between visits.

The patient will return for follow-up visit #3 for evaluation and management 8 weeks post-treatment intervention. At this visit, the following assessments will be completed:

- History and physical exam
- Patient self-assessment of both "general heel pain" and "first step pain" (VAS PROM)
- Patient self-assessment of foot function (FFI PROM)
- Dolorimeter readings of PPT # (pressure algometer)
- Heel tenderness score

Protocol version: 7

Review of the exercise diary

A new exercise diary will be given to the patient. The recommended exercises will be instructed again. Patients will be encouraged to bring the diary to their next visit. The patient will be called 1 last time to remind them of their exercise diary and encourage them to complete it.

The follow-up visit #4 will be the final study visit. This visit will occur 12 weeks post-treatment intervention. At this visit, the following assessments will be completed:

- History and physical exam
- Patient self-assessment of both "general heel pain" and "first step pain" (VAS PROM)
- Patient self-assessment of foot function (FFI PROM)
- Dolorimeter readings of PPT # (pressure algometer)
- Heel tenderness score
- Review of the exercise diary
- Final diagnostic musculoskeletal US (PF thickness and echogenicity; fat pad thickness)
- Exit survey

# **Evaluation Schedule Summary**

| | Screening | Injection | Week 2 | | Week 8 | Week 12 |
|---|---|---|---|---|---|---|
| | -42 to -1 | | +/- 3 | +/- 3 | +/- 3 | |
| Procedures | days | day 0 | days | days | days | +/- 3 days |
| Review Study Procedures, | | | | | | |
| Informed Consent, and Privacy | | | | | | |
| Authorization | X | Χ | | | | |
| Eligibility Criteria for Study | | | | | | |
| Entry | X | Х | | | | |
| Patient Demographics | X | | | | | |
| Patient Medical/Surgical | | | | | | |
| History | Х | Х | | | | |
| Height, Weight, and Vital Signs | Х | Х | Х | Х | Х | Х |
| Foot & Ankle Physical Exam | Х | Х | Х | Х | Х | Х |
| Presentation of Exercise | | | | | | |
| Therapy (targeted stretching and strengthening) | Х | x | x | х | x | x |
| Clinical Observation | X | X | , | X | X | X |
| X-ray of Affected Foot | Х | | | | | |
| Ultrasound of Affected Foot | Х | | | | | Х |
| Randomization | | Х | | | | |
| Study Therapeutic Treatment | | | | | | |
| Intervention (infracalcaneal | | | | | | |
| needle peppering injections) | | Х | | | | |
| Evaluation of Injection Site | | Х | Х | Х | Х | Х |

| Subject Self-Assessments - VAS PROM (for both general heel pain and first step pain) - FFI PROM | x | X | X | X | X | X |
|---|---|---|---|---|---|---|
| Exercise Diary & Instruction of the 3 Exercises | | x | X | X | X | Х |
| Foot Posture | Х | Х | | | | |
| Heel Pressure Threshold using Dolorimeter | x | X | Х | Х | X | Х |
| Heel Tenderness Score | Х | Х | Х | Х | Х | Х |
| Exit Survey | | | | | | Х |

<sup>\*</sup>Not on schedule: reminder phone call between study visits to encourage exercise diary completion and compliance.

# Outcome Measure(s)

Patient Assessments

- Heel Tenderness VAS PROM
- First Step Pain VAS PROM
- FFI PROM
- Exercise Diary
- Exit Survey at completion of study

#### Physician Assessments

- Baseline and subsequent foot and ankle physical exam, heel pressure threshold, and heel tenderness score
- X-ray and ultrasound imaging
  - Our research team will be the first to examine musculoskeletal ultrasound imaging obtained both before and after an infracalcaneal peppering injection in participants with chronic plantar fasciitis. Musculoskeletal ultrasound has become more established in the medical literature as a reliable objective measure of plantar fasciitis, with thickness measurements >4.0mm correlating with clinical symptoms (40). Musculoskeletal ultrasound's utility here would enable our investigators to assess for any quantifiable tissue changes associated with our intervention.

#### **Patient Retention**

Every effort will be made to retain patients in the study to ensure complete data collection. During the study consent process, potential study participants will be educated regarding the importance of full participation in all visits. Patients will be reminded of their upcoming appointment via phone call or email. Patients will also be reminded about their follow-up visits at all clinic visits.

Patient/study participant compensation will occur at certain study visits. Study participants will receive a paid total of \$100.00 if all scheduled study visits are completed.

| Study Visit #1 – injection day | \$20.00 |
|---|---|
| Study Visit #2 – 2 weeks post-treatment | No payment. Next payment at 4-week follow- |
| intervention | up study visit (visit #3). |
| Study Visit #3 – 4 weeks post-treatment | \$40.00 |
| intervention | |
| Study Visit #4 – 8 weeks post-treatment | No payment. Next payment at 12-week |
| intervention | follow-up study visit (visit #5). |
| Study Visit #5 – 12 weeks post-treatment | \$40.00 |
| intervention | |

### **Analytical Plan**

Results will be analyzed initially using descriptive statistics. Comparison between groups will be done using chi square tests for proportions, and t-tests or ANOVA procedures for continuous variables. Regression analysis will be performed to identify independent outcome predictors. Other inferential statistical analysis will be conducted as appropriate.

### **Human Subjects Protection**

All patients ages 18 years and up with a diagnosis of plantar heel pain will be screened for inclusion into the study. The study will be conducted in accordance with the current IRB-approved clinical protocol; ICH GCP Guidelines adopted by the FDA; relevant policies, requirements, and regulations of the clinical test site IRB; and applicable federal agencies.

Patients who meet the inclusion criteria will be asked to participate in the research study and provided ample time and encouragement to ask questions and discuss the study with others (medical providers, family, friends, etc.). A copy of the informed consent form will be provided to the patient. The study team will answer all questions.

Subjects may withdraw from the study at any time for any reason at their request. Otherwise, participants will be followed as per the protocol. Attempts will be made to collect clinical data from withdrawn subjects. There will be no replacement of subjects who withdraw from the study.

#### **Subject Recruitment Methods**

The study will recruit patients who present to the Atrium Health Wake Forest Baptist Department of Orthopaedic Surgery-Podiatry Services practice located in High Point, North Carolina with symptoms of plantar heel pain. In order to approach patients that have received care at this practice in the past, we will create an i2b2 query to result a list of patients seen by Dr. Jones and diagnosed with plantar fasciitis within the last 3 years (11/1/2020 – 11/1/2023). These patients will be contacted by the study coordinator to introduce the study, gauge their interest, and begin the pre-screening process if they opt in to doing so.

Additionally, the study will be listed on Be Involved and study flyers will be distributed and posted. A social media ad will also be distributed on Facebook and Instagram with information about the study and a link to the Be Involved web page. Interested potential subjects will be contacted via telephone or email and be asked to complete a pre-screening questionnaire. We will utilize a REDCap survey in instances where the potential subject prefers email communication to conduct the pre-screening questionnaire. Study flyers will have a QR code

available for interested individuals to scan and easily access the REDCap pre-screening questionnaire.

All completed questionnaires and personal identifying information collected via Be Involved, both for recruited subjects and those who have declined participation, will be kept securely by the select study personnel. This information will remain in a password protected file and only be accessed on a secure network.

### **Study Screening and Enrollment**

Potential study participants will be screened in the Orthopaedic Surgery-Podiatry Services Practice. Patients with plantar heel pain who meet the study inclusion criteria will be told about the study and will be asked if they would like to participate. The study will be described, and the requirements for study participation will be explained. Potential study participants will be encouraged to ask questions about the study and to find out what is involved in study participation. Patients who agree to participate will be asked to provide informed consent. No study related procedures will occur until after the informed consent is obtained. Following completion of informed consent, the study procedures will begin.

## **Informed Consent**

Signed informed consent will be obtained from each subject in the privacy of a closed clinical examination room. A study team member will discuss the study with patients who meet study entry criteria and will obtain consent while the patients are in the clinic following their visit. Each study participant will receive a copy of the signed informed consent form.

## **Confidentiality and Privacy**

Confidentiality will be protected by collecting only information needed to assess study outcomes, fully minimizing the collection of any information that could directly identify subjects and maintaining all study information in a secure manner. To help ensure subject privacy and confidentiality, only a unique study identifier will appear on the data collection form. Any collected patient identifying information corresponding to the unique study identifier will be maintained on a linkage file and stored separately from the data. The linkage file will be kept secure, with access limited to designated study personnel. Following data collection, subject identifying information will be destroyed six years after closure of the study by shredding any paper documents and deleting information from computer files, consistent with data validation and study design, producing an anonymous analytical data set. Data access will be limited to study staff. Data and records will be kept locked and secured, with computer data being password protected. No reference to any individual participant will appear in reports, presentations, or publications that may arise from the study.

## **Data and Safety Monitoring**

The principal investigator will be responsible for the overall monitoring of the data and safety of study participants. The principal investigator will be assisted by other members of the study staff.

#### Reporting of Unanticipated Problems, Adverse Events or Deviations

Protocol version: 7

Any unanticipated problems, serious and unexpected adverse events, deviations or protocol changes will be promptly reported by the principal investigator or designated member of the research team to the IRB and sponsor or appropriate government agency if appropriate.

#### References

- 1. Riddle DL, Schappert SM. Volume of ambulatory care visits and patterns of care for patients diagnosed with plantar fasciitis: a national study of medical doctors. Foot Ankle Int. 2004 May;25(5):303-10. doi: 10.1177/107110070402500505. PMID: 15134610.
- 2. Tong KB, Furia J. Economic burden of plantar fasciitis treatment in the United States. Am J Orthop (Belle Mead NJ). 2010 May;39(5):227-31. PMID: 20567740.
- 3. Stecco C, Corradin M, Macchi V, Morra A, Porzionato A, Biz C, De Caro R. Plantar fascia anatomy and its relationship with Achilles tendon and paratenon. J Anat. 2013 Dec;223(6):665-76. doi: 10.1111/joa.12111. Epub 2013 Sep 12. PMID: 24028383; PMCID: PMC3842207.
- 4. HICKS JH. The mechanics of the foot. I. The joints. J Anat. 1953 Oct;87(4):345-57. PMID: 13117752; PMCID: PMC1244617.
- Wearing SC, Smeathers JE, Urry SR, Hennig EM, Hills AP. The pathomechanics of plantar fasciitis. Sports Med. 2006;36(7):585-611. doi: 10.2165/00007256-200636070-00004. PMID: 16796396.
- van Leeuwen KD, Rogers J, Winzenberg T, van Middelkoop M. Higher body mass index is associated with plantar fasciopathy/'plantar fasciitis': systematic review and metaanalysis of various clinical and imaging risk factors. Br J Sports Med. 2016 Aug;50(16):972-81. doi: 10.1136/bjsports-2015-094695. Epub 2015 Dec 7. PMID: 26644427.
- 7. Bolívar YA, Munuera PV, Padillo JP. Relationship between tightness of the posterior muscles of the lower limb and plantar fasciitis. Foot Ankle Int. 2013 Jan;34(1):42-8. doi: 10.1177/1071100712459173. PMID: 23386760.
- 8. Buchbinder R. Clinical practice. Plantar fasciitis. N Engl J Med. 2004 May 20;350(21):2159-66. doi: 10.1056/NEJMcp032745. PMID: 15152061.
- 9. Cotchett M, Munteanu SE, Landorf KB. Depression, Anxiety, and Stress in People With and Without Plantar Heel Pain. Foot Ankle Int. 2016 Aug;37(8):816-21. doi: 10.1177/1071100716646630. Epub 2016 May 2. PMID: 27137796.
- 10. Irving DB, Cook JL, Young MA, Menz HB. Impact of chronic plantar heel pain on health-related quality of life. J Am Podiatr Med Assoc. 2008 Jul-Aug;98(4):283-9. doi: 10.7547/0980283. PMID: 18685048.
- 11. Schneider HP, Baca JM, Carpenter BB, Dayton PD, Fleischer AE, Sachs BD. American College of Foot and Ankle Surgeons Clinical Consensus Statement: Diagnosis and Treatment of Adult Acquired Infracalcaneal Heel Pain. J Foot Ankle Surg. 2018 Mar-Apr;57(2):370-381. doi: 10.1053/j.jfas.2017.10.018. Epub 2017 Dec 25. PMID: 29284574.
- 12. Goff JD, Crawford R. Diagnosis and treatment of plantar fasciitis. Am Fam Physician. 2011 Sep 15;84(6):676-82. PMID: 21916393.
- 13. Hansen L, Krogh TP, Ellingsen T, Bolvig L, Fredberg U. Long-Term Prognosis of Plantar Fasciitis: A 5- to 15-Year Follow-up Study of 174 Patients With Ultrasound Examination. Orthop J Sports Med. 2018 Mar 6;6(3):2325967118757983. doi: 10.1177/2325967118757983. PMID: 29536022; PMCID: PMC5844527.

- 14. AOFAS Choosing Wisely. <a href="https://www.choosingwisely.org/wp-content/uploads/2015/11/AOFAS Treating-plantar-fasciitis.pdf">https://www.choosingwisely.org/wp-content/uploads/2015/11/AOFAS Treating-plantar-fasciitis.pdf</a>. Published 2015. Accessed November 20, 2022.
- 15. Buchbinder, R., Isaac, Z. (2022). Plantar Fasciitis. *UpToDate*. Retrieved November 20, 2022 from <a href="https://www.uptodate.com/contents/plantarfasciitis?search=plantar%20fasciitis&source=search=result&selectedTitle=1~40&usage\_type=default&display\_rank=1">https://www.uptodate.com/contents/plantarfasciitis?search=plantar%20fasciitis&source=search=result&selectedTitle=1~40&usage\_type=default&display\_rank=1</a>
- 16. David JA, Sankarapandian V, Christopher PR, Chatterjee A, Macaden AS. Injected corticosteroids for treating plantar heel pain in adults. Cochrane Database Syst Rev. 2017 Jun 11;6(6):CD009348. doi: 10.1002/14651858.CD009348.pub2. PMID: 28602048; PMCID: PMC6481652.
- 17. BLOCKEY NJ. The painful heel; a controlled trial of the value of hydrocortisone. Br Med J. 1956 Jun 2;1(4978):1277-8. doi: 10.1136/bmj.1.4978.1277. PMID: 13316131; PMCID: PMC1979664.
- 18. Fadale PD, Wiggins ME. Corticosteroid Injections: Their Use and Abuse. J Am Acad Orthop Surg. 1994 May;2(3):133-140. doi: 10.5435/00124635-199405000-00001. PMID: 10709001.
- 19. Schneider HP, Baca JM, Carpenter BB, Dayton PD, Fleischer AE, Sachs BD. American College of Foot and Ankle Surgeons Clinical Consensus Statement: Diagnosis and Treatment of Adult Acquired Infracalcaneal Heel Pain. J Foot Ankle Surg. 2018 Mar-Apr;57(2):370-381. doi: 10.1053/j.jfas.2017.10.018. Epub 2017 Dec 25. PMID: 29284574.
- 20. D'Ambrosia RD. Conservative management of metatarsal and heel pain in the adult foot. Orthopedics. 1987 Jan;10(1):137-42. doi: 10.3928/0147-7447-19870101-25. PMID: 3809011.
- 21. Lee HS, Choi YR, Kim SW, Lee JY, Seo JH, Jeong JJ. Risk factors affecting chronic rupture of the plantar fascia. Foot Ankle Int. 2014 Mar;35(3):258-63. doi: 10.1177/1071100713514564. Epub 2013 Nov 25. PMID: 24275488.
- 22. Rhim HC, Kwon J, Park J, Borg-Stein J, Tenforde AS. A Systematic Review of Systematic Reviews on the Epidemiology, Evaluation, and Treatment of Plantar Fasciitis. Life (Basel). 2021 Nov 24;11(12):1287. doi: 10.3390/life11121287. PMID: 34947818: PMCID: PMC8705263.
- 23. Berbrayer D, Fredericson M. Update on evidence-based treatments for plantar fasciopathy. PM R. 2014 Feb;6(2):159-69. doi: 10.1016/j.pmrj.2013.08.609. Epub 2013 Dec 21. PMID: 24365781.
- 24. Lemont H, Ammirati KM, Usen N. Plantar fasciitis: a degenerative process (fasciosis) without inflammation. J Am Podiatr Med Assoc. 2003 May-Jun;93(3):234-7. doi: 10.7547/87507315-93-3-234. PMID: 12756315.
- 25. Trojian T, Tucker AK. Plantar Fasciitis. Am Fam Physician. 2019 Jun 15;99(12):744-750. PMID: 31194492.
- 26. Riel H, Vicenzino B, Jensen MB, Olesen JL, Holden S, Rathleff MS. The effect of isometric exercise on pain in individuals with plantar fasciopathy: A randomized crossover trial. Scand J Med Sci Sports. 2018 Dec;28(12):2643-2650. doi: 10.1111/sms.13296. Epub 2018 Oct 1. PMID: 30203866.
- 27. Rathleff MS, Mølgaard CM, Fredberg U, Kaalund S, Andersen KB, Jensen TT, Aaskov S, Olesen JL. High-load strength training improves outcome in patients with plantar fasciitis: A randomized controlled trial with 12-month follow-up. Scand J Med Sci Sports.

- 2015 Jun;25(3):e292-300. doi: 10.1111/sms.12313. Epub 2014 Aug 21. PMID: 25145882.
- 28. Vajapey S, Ghenbot S, Baria MR, Magnussen RA, Vasileff WK. Utility of Percutaneous Ultrasonic Tenotomy for Tendinopathies: A Systematic Review. Sports Health. 2021 May-Jun;13(3):258-264. doi: 10.1177/1941738120951764. Epub 2020 Nov 30. PMID: 33252310; PMCID: PMC8083144.
- Prakash YR, Dhanda A, Yallapur KL, Inamdar SS, Darshan GT, Ramakrishna M. Peppering versus Single Injection Technique in Tennis Elbow - A Prospective Comparative Study. Malays Orthop J. 2022 Mar;16(1):91-96. doi: 10.5704/MOJ.2203.013. PMID: 35519523; PMCID: PMC9017907.
- 30. PRUCE AM, MILLER JA Jr, BERGER IR. ANATOMIC LANDMARKS IN JOINT PARACENTESIS. Clin Symp. 1964 Jan-Mar;16:19-30. PMID: 14111853.
- 31. Chiavaras MM, Jacobson JA. Ultrasound-guided tendon fenestration. Semin Musculoskelet Radiol. 2013 Feb;17(1):85-90. doi: 10.1055/s-0033-1333942. Epub 2013 Mar 13. PMID: 23487340.
- 32. Altay T, Günal I, Oztürk H. Local injection treatment for lateral epicondylitis. Clin Orthop Relat Res. 2002 May;(398):127-30. PMID: 11964641.
- 33. (29) Prakash YR, Dhanda A, Yallapur KL, Inamdar SS, Darshan GT, Ramakrishna M. Peppering versus Single Injection Technique in Tennis Elbow A Prospective Comparative Study. Malays Orthop J. 2022 Mar;16(1):91-96. doi: 10.5704/MOJ.2203.013. PMID: 35519523; PMCID: PMC9017907.
- 34. Okçu G, Erkan S, Sentürk M, Ozalp RT, Yercan HS. Evaluation of injection techniques in the treatment of lateral epicondylitis: a prospective randomized clinical trial. Acta Orthop Traumatol Turc. 2012;46(1):26-9. doi: 10.3944/aott.2012.2577. PMID: 22441448.
- 35. Kiter E, Celikbas E, Akkaya S, Demirkan F, Kiliç BA. Comparison of injection modalities in the treatment of plantar heel pain: a randomized controlled trial. J Am Podiatr Med Assoc. 2006 Jul-Aug;96(4):293-6. doi: 10.7547/0960293. PMID: 16868321.
- 36. Kalaci A, Cakici H, Hapa O, Yanat AN, Dogramaci Y, Sevinç TT. Treatment of plantar fasciitis using four different local injection modalities: a randomized prospective clinical trial. J Am Podiatr Med Assoc. 2009 Mar-Apr;99(2):108-13. doi: 10.7547/0980108. PMID: 19299346.
- 37. Dogramaci Y, Kalaci A, Savaş N, Duman IG, Yanat AN. Treatment of lateral epicondilitis using three different local injection modalities: a randomized prospective clinical trial. Arch Orthop Trauma Surg. 2009 Oct;129(10):1409-14. doi: 10.1007/s00402-009-0832-x. Epub 2009 Feb 14. PMID: 19219442.
- 38. Ball EM, McKeeman HM, Patterson C, Burns J, Yau WH, Moore OA, Benson C, Foo J, Wright GD, Taggart AJ. Steroid injection for inferior heel pain: a randomised controlled trial. Ann Rheum Dis. 2013 Jun;72(6):996-1002. doi: 10.1136/annrheumdis-2012-201508. Epub 2012 Jun 27. PMID: 22739993.
- 39. Crawford F, Atkins D, Young P, Edwards J. Steroid injection for heel pain: evidence of short-term effectiveness. A randomized controlled trial. Rheumatology (Oxford). 1999 Oct;38(10):974-7. doi: 10.1093/rheumatology/38.10.974. PMID: 10534548.
- 40. Salehi S, Shadmehr A, Olyaei G, Bashardoust Tajali S, Mir SM, Sobhani V. Ultrasonographic measurements of plantar fascia thickness and echogenicity in individuals with and without plantar fasciitis: Reliability and group differences. Foot

(Edinb). 2021 Dec;49:101849. doi: 10.1016/j.foot.2021.101849. Epub 2021 Jul 8. PMID: 34597921.

# **Appendix**

- 1. Data Collection Sheet
- 2. VAS PROM
- 3. FFI PROM
- 4. Exercise Diary
- 5. Exit Survey